CLINICAL TRIAL: NCT01538212
Title: Retrospective Cohort Study Of The Efficacy Of Axona® (Medium Chain Triglycerides) In Patients With Alzheimer's Disease
Acronym: ACT
Status: Completed | Type: Observational
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Other Study IDs: AX-11-009
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; retrospective; Axona
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This evaluation of the efficacy and safety of AXONA will be a chart review carried out at 16 practices in which AXONA has been prescribed for the treatment of patients with mild-to-moderate AD. Efficacy of AXONA will be assessed by comparison of patient status before and after initiation of treatment.

DETAILED DESCRIPTION:
The primary objective is to assess the efficacy of AXONA (medium chain triglycerides [MCTs]) when used alone or in combination with other agents in patients with mild-to-moderate Alzheimer's disease (AD) in routine clinical practice.

ELIGIBILITY:
Patient Inclusion Criteria:

* Male or female outpatients aged ≥ 50 years with a diagnosis of probable AD of mild-to-moderate severity
* MMSE score between 14 and 24 inclusive at the initiation of AXONA treatment (if available)
* Has received Axona for a duration of ≥ 6 months

Caregiver Inclusion Criteria (if applicable):

* Must be at least 21 years of age, has been the primary caregiver since prior to the initiation of Axona, provides at least 4 hours of supervision or direct assistance per day for the patient and is able to perform assessments.

Patient Exclusion Criteria:

* MMSE score < 14 at the time when AXONA treatment was initiated
* Presence of co-morbid disease known to adversely impact cognitive function (e.g., Parkinson's disease, history of cerebral infarcts, dementia with Lewy bodies)
* Vascular dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with a diagnosis of mild-to-moderate AD who have been treated with AXONA for ≥ 6 months and whose medical record includes an evaluation within 3 months prior to initiation of treatment and at least one evaluation while receiving AXONA.
  Potential for intentional inclusion in the study will be determined on the basis of prescribing data and physicians will be contacted. For Neurology and Psychiatry practices agreeing to participate, all charts meeting the above criteria and for which patients/caregivers give consent will be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Physician's Overall Assessment of Patient Status at the beginning of Axona treatment and the most recent assessment | 6 months post the start date of Axona

SECONDARY OUTCOMES:
Changes from baseline in patient's living situation | 6 months post the start date of Axona
Changes from baseline in patient's medications for the treatment of AD | 6 months post the start date of Axona
Changes from baseline in patient's medications for psychiatric conditions related to AD | 6 months post the start date of Axona
Changes from baseline in patient's memory and ability to carry out instrumental activities of daily living as assessed by caregivers | 6 months post the start date of Axona
Adverse events assessed by physician's as being possibly associated with the use of Axona | 6 months post the start date of Axona

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T Henderson, PhD, Study Director — Cerecin